CLINICAL TRIAL: NCT03217734
Title: MAP Study (Methotrexate and Adalimumab in Psoriasis): Adalimumab vs. Combination Adalimumab and Methotrexate in Psoriasis: Efficacy and Anti-Adalimumab Antibody Formation
Brief Title: MAP Study: Methotrexate and Adalimumab in Psoriasis
Acronym: MAP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jeffrey J Crowley MD (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey J Crowley MD, Jeffrey J Crowley, MD, Prinicipal Investigator, Bakersfield Dermatology & Skin Cancer Medical Group
Organization: Bakersfield Dermatology & Skin Cancer Medical Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A16-241
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ADA and Placebo (Placebo Comparator): Adalimumab 40 mg, Subcutaneous, Bi-Weekly, 16 Weeks Placebo, Tablet, Oral, Weekly, 16 Weeks
  Interventions: Biological: Adalimumab; Drug: Placebo
- ADA and MTX (Active Comparator): Adalimumab 40 mg, Subcutaneous, Bi-Weekly, 16 Weeks Methotrexate, 2.5 mg Tablet, 10 mg Weekly, Oral, 16 Weeks
  Interventions: Biological: Adalimumab; Drug: Methotrexate

INTERVENTIONS:
Biological: Adalimumab — Subcutaneous Injection
  Other Names: Humira
Drug: Methotrexate — Oral Tablet
  Other Names: MTX
  Arms: ADA and MTX
Drug: Placebo — Oral Tablet
  Arms: ADA and Placebo

SUMMARY:
Assess the efficacy and safety of ADA compared to ADA/MTX in patient with Psoriasis. Compare Anti-ADA antibody formation and serum ADA levels in patients on ADA compared with those on combination ADA and MTX.

DETAILED DESCRIPTION:
Assess the efficacy and safety of ADA compared to ADA/MTX in patients with psoriasis. Many studies of ADA in rheumatoid and psoriatic arthritis have allowed patients on stable doses of MTX to continue on MTX while being treated with ADA. There has been no prospective trial of MTX and ADA concomitantly in psoriasis. Safety of ADA monotherapy vs. combination ADA/MTX will be compared.

Compare anti-ADA antibody formation and serum ADA levels in patients on ADA compared with those on combination ADA and MTX. ADA is a fully human monoclonal antibody to TNF-a. More recent advances in detection of ADA antibodies have shown that many patients develop antibodies to ADA while on treatment and some of these antibodies are neutralizing. The presence of anti-ADA antibodies has been correlated with loss of therapeutic response in many disease states.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult (≥ 18yrs) with a diagnosis of moderate to severe plaque psoriasis
2. Subject must have ≥ 10% body surface area involvement
3. Subject must have psoriasis area and severity index (PASI) ≥12
4. Subject has stable psoriasis of at least six months' duration
5. Male subjects must agree to use a reliable form of birth control during the study and for 180 days after the last dose of study drug. Male subjects must not donate sperm during the study or for 180 days after the last dose of study drug. If female, subject is either not of childbearing potential (postmenopausal for at least 1 year or surgically sterile) or is of childbearing potential and is using approved method of birth control throughout study and for 180 days after last dose of study drug. Approved methods of birth control include the following:

   1. Condoms, sponge, foams, jellies, diaphragm, or intrauterine device (IUD)
   2. Hormonal contraceptives for 90 days prior to study drug administration
   3. A vasectomized partner
6. Subject has negative PPD tuberculosis skin test at screening assessment.
7. Subject must be able and willing to provide written informed consent and comply with requirements of this study protocol.

Exclusion Criteria

1. Diagnosis or presence of guttate, erythrodermic or pustular psoriasis
2. Any previous exposure to ADA including biosimilar ADA
3. Moderate to high strength topical steroids (class 4 or greater) or Vitamin D analogues within one week of study entry
4. Oral systemic therapy (methotrexate, cyclosporine, apremilast, acitretin) within 8 weeks of study entry
5. Previous intolerance or adverse reaction to MTX
6. Phototherapy of any type within 4 weeks of study entry (narrowband UVB, psoralen-UVA, 308 nM LASER, commercial tanning units)
7. IL-12/23 inhibitors (ustekinumab) and any IL-23 inhibitor (guselkumab, tildrakizumab, risankizumab) within 12 weeks of baseline
8. Other biologic agents within 8 weeks of study entry
9. History of chronic liver disease, hepatitis, or alcohol abuse
10. Chronic use of any concomitant medication which has a significant potential for interaction with MTX (e.g. sulfa antibiotics, chronic non-steroidal anti-inflammatory (NSAID) use)
11. History of tuberculosis, opportunistic infections, or any active infection at screening
12. Elevated liver enzymes (AST, ALT, ≥1.5 times normal at screening)
13. Serum creatinine ≥1.5 (at screening)
14. Any other laboratory abnormality that would pose a concern for the investigator
15. Daily alcohol use or consumption of more than four alcoholic drinks (4 ounces) in one 24 hour period
16. Patients who test positive for hepatitis B or C exposure (previous vaccination to Hepatitis B is allowed)
17. Cancer within the last five years is exclusionary with the exception of treated cutaneous basal cell carcinoma or squamous cell carcinoma or low-grade cervical intraepithelial neoplasia.
18. Any patient that is deemed by the investigator to be at a safety risk for the intervention in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
PASI Change | 16 weeks
  Mean percent change in PASI from 16 Weeks to Baseline

SECONDARY OUTCOMES:
ADA/Anti ADA Antibodies | 16 weeks
  Antibodies to Adalimumab at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Crowley, MD, Study Director — Bakersfield Dermatology and Skin Cancer Medical Group
Locations (4):
- United States (4):
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Clinical Science Institute, Santa Monica, California
  - DermAssociates, PC, Rockville, Maryland
  - Modern Research Associates, PLLC, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No